CLINICAL TRIAL: NCT05078736
Title: Effects of Moderate Intensity Intermittent Training Versus Continuous Training on Indices of Cardio-metabolic Health in Women With Hyperlipidemia
Brief Title: Effects of Moderate Intensity Intermittent and Moderate Intensity Continuous Training on Hyperlipdemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/Lhr/0409 Shama
Record Dates: First submitted 2021-08-27; First posted 2021-10-14 (Actual); Last update posted 2022-01-04 (Actual); Status verified 2022-01

CONDITIONS: Hyperlipidemias
Keywords: Cholesterol; Hyperlipidemia; MICT; MIIT
MeSH Terms: conditions — Hyperlipidemias

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- moderate intensity intermittent training (Experimental): baseline physical therapy treatment along with moderate intensity intermittent training
  Interventions: Other: Moderate intensity intermittent training
- moderate intensity continuous training (Experimental): baseline physical therapy treatment along with moderate intensity continuous training
  Interventions: Other: Moderate intensity continuous training

INTERVENTIONS:
Other: Moderate intensity intermittent training — In group A participants will receive moderate intensity intermittent training including running of 5 km with 1-min at 70% of maximal aerobic speed with interval of 1-min passive recovery, exercises will be performed by gym trainer for 5 weeks including 3 days/week
  Arms: moderate intensity intermittent training
Other: Moderate intensity continuous training — In group B participants will receive moderate intensity continuous training ran continuously the same 5 km at 70% of maximal aerobic speed, exercises will be performed by gym trainer for 5 weeks including 3 days/week.
  Arms: moderate intensity continuous training

SUMMARY:
This project will be a Randomized control trial conducted to check the effects of moderate intensity intermittent training versus moderate intensity continuous training on indices of cardio-metabolic health in women with hyperlipidemia, duration will be of 5 weeks, purposive sampling data technique, will be done, subject following eligibility criteria from milestone gym Sialkot, will randomly allocated in two groups via lottery method, baseline assessment will be done, Group A participants will receive baseline treatment along with moderate intensity intermittent training, and Group B participants will receive baseline treatment along with moderate intensity continuous training. Pre and post intervention assessment will include lipid profile test and Vo2 max rating of perceived exertion (RPE), and post data will be analyzed by using SPSS version 25.

DETAILED DESCRIPTION:
Hyperlipidemia is a condition with high levels of fat in the blood, such as cholesterol and triglycerides. Hyperlipidemia is most commonly associated with high-fat diets, sedentary lifestyle, obesity and diabetes. The aim of the current study is to find the effectiveness of moderate intensity intermittent training and moderate intensity continuous training in women with hyperlipidemia. It will be a Randomized control trial and screening will be done as per the inclusion criteria of women having 30-40 years of age with hyperlipidemia. Participants with the history of any serious cardiac condition, musculoskeletal injury, and any type of systemic issue will be excluded.

Participants will be randomly allocated into two groups, Group A will receive moderate intensity intermittent training consist of running for 5 km with 1-min at 70% of maximal aerobic speed with interval of 1-min passive recovery and Group B will receive moderate intensity continuous training consist of running continuously for 5 km at 70% of maximal aerobic speed for 5 weeks including exercise training of 3 days/week. Participants in both groups will be assessed with Lipid profile (fasting triglycerides, High Density Lipoproteins, Low density Lipoproteins) before and after the intervention.

VO2 max, rating of perceived exertion (RPE) Step Test: The step test is designed to measure a person's aerobic fitness. Participants step up and down, on and off an aerobic- type step for three minutes to increase heart rate and evaluate the heart's recovery rate during the minute immediately following the step test exercise.

Modified Borg scale: MBS is a 0-10 rated numerical score used to measure dyspnea as reported by the patient during submaximal exercise and is routinely administrated during six-minute walk testing.

ELIGIBILITY:
Inclusion Criteria:

* Women.
* Age 30-40 years.
* Hyperlipidemia

Exclusion Criteria:

* With another serious cardiac condition.
* With any musculoskeletal injury.
* With any systematic condition.

Ages: 30 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 20 (Actual)
Dates: Start 2021-08-30 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Lipid profile | 5 weeks
  Lipid profile (fasting triglycerides, HDL, LDL) will be done through blood samples of the participants.
Step Test: | 5th Week
  The step test is designed to measure a person's aerobic fitness. Participants step up and down, on and off an aerobic- type step for three minutes to increase heart rate and evaluate the heart's and evaluate the heart's recovery rate during the minute immediately following the step test exercise.
Modified Borg scale | 5th Week
  MBS is a 0-10 rated numerical score used to measure dyspnea as reported by the patient during submaximal exercise and is routinely administrated during six-minute walk testing.

CONTACTS AND LOCATIONS:
Overall Officials: Syed Shakil Ur Rehman, Principal Investigator — Riphah International University
Locations (1):
- Sialkot, Milestone gym, Sialkot, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nirosha K, Divya M, Vamsi S, Sadiq M. A review on hyperlipidemia. International Journal of Novel Trends in PharmaceuticalSciences. 2014;4(5):81-92
- [Background] Fung M, Hill J, Cook D, Frohlich J. Case series of type III hyperlipoproteinemia in children. BMJ Case Rep. 2011 Jun 9;2011:bcr0220113895. doi: 10.1136/bcr.02.2011.3895. PMID 22691586
- [Background] Kinoshita M, Yokote K, Arai H, Iida M, Ishigaki Y, Ishibashi S, Umemoto S, Egusa G, Ohmura H, Okamura T, Kihara S, Koba S, Saito I, Shoji T, Daida H, Tsukamoto K, Deguchi J, Dohi S, Dobashi K, Hamaguchi H, Hara M, Hiro T, Biro S, Fujioka Y, Maruyama C, Miyamoto Y, Murakami Y, Yokode M, Yoshida H, Rakugi H, Wakatsuki A, Yamashita S; Committee for Epidemiology and Clinical Management of Atherosclerosis. Japan Atherosclerosis Society (JAS) Guidelines for Prevention of Atherosclerotic Cardiovascular Diseases 2017. J Atheroscler Thromb. 2018 Sep 1;25(9):846-984. doi: 10.5551/jat.GL2017. Epub 2018 Aug 22. No abstract available. PMID 30135334
- [Background] Zhang ZH, Wei F, Vaziri ND, Cheng XL, Bai X, Lin RC, Zhao YY. Metabolomics insights into chronic kidney disease and modulatory effect of rhubarb against tubulointerstitial fibrosis. Sci Rep. 2015 Sep 28;5:14472. doi: 10.1038/srep14472. PMID 26412413
- [Background] Alvarez Ramirez AA, Pelaez JL, Bermudez IM, Gordon Botero JY. Prevalence of hyperlipidemia and its associated factors in university students in Colombia. Heliyon. 2020 Nov 3;6(11):e05417. doi: 10.1016/j.heliyon.2020.e05417. eCollection 2020 Nov. PMID 33195846
- [Background] Abid N, Khan SA, Taseer I. Frequency of hyperlipidemia in patients presenting with ischemic stroke. Pak J Med Health Sci. 2012;6(2):423-28
- [Background] Nelson RH. Hyperlipidemia as a risk factor for cardiovascular disease. Prim Care. 2013 Mar;40(1):195-211. doi: 10.1016/j.pop.2012.11.003. Epub 2012 Dec 4. PMID 23402469
- [Background] Caballero B, Trugo LC, Finglas PM. Encyclopedia of food sciences and nutrition: Academic; 2003
- [Background] Pramparo P, Boissonnet C, Schargrodsky H. Evaluation of Cardiovascular Risk in Seven Cities in Latin America: The Main Conclusions. Argentine Journal of Cardiology.79(4):368-70
- [Background] Lira FS, Antunes BM, Figueiredo C, Campos EZ, Panissa VLG, St-Pierre DH, Lavoie JM, Magri-Tomaz L. Impact of 5-week high-intensity interval training on indices of cardio metabolic health in men. Diabetes Metab Syndr. 2019 Mar-Apr;13(2):1359-1364. doi: 10.1016/j.dsx.2019.02.006. Epub 2019 Feb 5. PMID 31336492
- [Background] Alansare A, Alford K, Lee S, Church T, Jung HC. The Effects of High-Intensity Interval Training vs. Moderate-Intensity Continuous Training on Heart Rate Variability in Physically Inactive Adults. Int J Environ Res Public Health. 2018 Jul 17;15(7):1508. doi: 10.3390/ijerph15071508. PMID 30018242
- [Background] Khan SU, Khan MZ, Raghu Subramanian C, Riaz H, Khan MU, Lone AN, Khan MS, Benson EM, Alkhouli M, Blaha MJ, Blumenthal RS, Gulati M, Michos ED. Participation of Women and Older Participants in Randomized Clinical Trials of Lipid-Lowering Therapies: A Systematic Review. JAMA Netw Open. 2020 May 1;3(5):e205202. doi: 10.1001/jamanetworkopen.2020.5202. PMID 32437574